CLINICAL TRIAL: NCT07106489
Title: Effect of Beetroot Extract Supplementation on the Athletic Performance of Trained Rugby Athletes
Brief Title: Effect of Beetroot Nitrates on Different Physical Skills in Colombian Rugby Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional de Colombia (Other)
Responsible Party: Principal Investigator, Ligia Stella Guerrero Orjuela, PhD. MSc. ND. Professor, Universidad Nacional de Colombia
Allocation: Non-Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 65891
Record Dates: First submitted 2025-07-22; First posted 2025-08-06 (Actual); Results first posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-06

CONDITIONS: Athletic Performance
Keywords: Beetroot; Nitrates; Sports; Sports Nutrition Science

STUDY DESIGN:
Intervention Model Description: The research was a quasi-experimental study using a non-randomized controlled crossover trial, minimizing the effects associated with individual athlete patterns, with each participant acting as their own control. Participants were double-blinded, dividing them into two groups. The researcher prepared placebo and beetroot waffles.
Who Masked: Participant, Care Provider, Investigator
Masking Description: A person external to the study was tasked with providing a compound to each group and ensuring they were exchanged during the second sample collection, ensuring that both groups received both compounds (the placebo and nitrates) at the end of the study. The professional who performed the physical tests was also blinded throughout the study. Thus, participants knew they would receive a placebo and beetroot, but they were not aware of the order in which they were given the compound.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo-Beetroot (Other): The group receives the placebo the first week and the following week they receive the beetroot
  Interventions: Other: beetroot juice - Placebo; Other: 40 meters sprint; Other: Fitness test by bronco test; Other: Maximal strength; Other: Borg scale
- Beetroot-Placebo (Other): The group receives the beetroot the first week and the following week receives the placebo.
  Interventions: Other: beetroot juice - Placebo; Other: 40 meters sprint; Other: Fitness test by bronco test; Other: Maximal strength; Other: Borg scale

INTERVENTIONS:
Other: beetroot juice - Placebo — Participants receive the beetroot and placebo in the form of waffles to ensure the study is blinded, as the 6 mmol of nitrates used require a high concentration of beetroot, which is masked by the waffle ingredients and food coloring.
Other: 40 meters sprint — The participant performs a race at maximum speed with two attempts, times are taken at 10, 30 and 40 meters, to evaluate acceleration and speed, the attempt with the shortest times is the one taken for the research.
Other: Fitness test by bronco test — The participant runs a distance of 20, 40, and 60 meters, back and forth, 5 times at maximum speed. The variable to be measured is the total time taken to complete the test.
Other: Maximal strength — Each participant performs squats and bench press to evaluate lower-body and upper-body maximal strength, thus identifying their maximum strength taken per kilogram lifted.
Other: Borg scale — At the end of the tests, each participant is asked to evaluate their perception of fatigue by giving a number between 1 and 10, with 1 being the lowest level of fatigue and 10 being the highest.

SUMMARY:
Beetroot is a source of nitrates, which have demonstrated various positive effects in sports, with little evidence in intermittent sports such as ball sports (including rugby). Therefore, the study's hypothesis is that it may also have an effect in these sports. For this purpose, a beetroot extract was used, a product approved by the Colombian institution in charge of product approval and registration in Colombia, the National Institute for Food and Drug Surveillance (INVIMA). This was done to determine whether it has any effect on various physical abilities required for rugby, such as speed, acceleration, strength, and fatigue perception.

DETAILED DESCRIPTION:
Currently, nitrates (from beet juices or extracts) have gained relevance due to their vasodilatory effect, which has contributed to improving athletic performance. Their use has been studied mainly in continuous sports such as swimming, cycling, athletics, etc. However, research in intermittent sports (such as ball or combat sports) is limited and inconclusive, so further research is needed on their use and effect in these sports. Therefore, the study seeks to investigate the effect of administering beet extract for three consecutive days in rugby athletes, evaluating its effect on various physical capacities required for the specific sport, such as acceleration, speed, strength, and fitness. Due to the small number of participants, a randomization process is not possible. A representative sample of 44 is required, but only 10 are interested in participating. Therefore, the sample will be selected based on the number of people willing to participate (convenience sampling) and meeting the defined inclusion and exclusion criteria. Each athlete is subsequently characterized and evaluated by the nutritionist, who provides instructions on how to avoid consuming foods or substances that could affect the study. They will be provided with the necessary substrates three days before the physical tests, with one group receiving the beetroot substrate and the other a placebo. The following week, the groups will be double-blinded. The physical tests will be performed by a professional physiotherapist, who will apply the test protocol and use a Borg scale to assess perceived exertion. Finally, a descriptive and exploratory analysis will be performed on the collected data, using univariate tests for the mean (Student's t-test) or Wilcoxon tests, depending on the type of variable (continuous or ordinal), with a 95% confidence level. To measure the magnitude of the treatment effect on each measured variable, Cohen's d statistic will be used for those variables that required a t-test.

ELIGIBILITY:
Inclusion Criteria:

* Belong to one of the two Rugby Clubs invited to participate
* Legal age
* Have trained/played rugby for more than 6 months.

Exclusion Criteria:

* Have had a sports injury in the last 6 months or during the study
* Use of nutritional supplements during the study.
* Use of mouthwash during the study.
* Have health conditions that require specific medical treatment.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-03-05 (Actual); Study Completion 2025-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ligia S Guerrero, PhD. MSc. ND, Study Director — Universidad Nacional de Colombia
Locations (1):
- Universidad Nacional de Colombia, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: Yes
The study is expected to be written and submitted to peer-reviewed, indexed journals in areas such as nutrition, exercise physiology, and public health.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Beginning once the scientific article is been accepted and with no end date
Access Criteria: The criteria given by the chosen journal will be taken into account

REFERENCES:
- [Background] Thompson C, Vanhatalo A, Jell H, Fulford J, Carter J, Nyman L, Bailey SJ, Jones AM. Dietary nitrate supplementation improves sprint and high-intensity intermittent running performance. Nitric Oxide. 2016 Dec 30;61:55-61. doi: 10.1016/j.niox.2016.10.006. Epub 2016 Oct 21. PMID 27777094
- [Background] Tan R, Pennell A, Karl ST, Cass JK, Go K, Clifford T, Bailey SJ, Perkins Storm C. Effects of Dietary Nitrate Supplementation on Back Squat and Bench Press Performance: A Systematic Review and Meta-Analysis. Nutrients. 2023 May 27;15(11):2493. doi: 10.3390/nu15112493. PMID 37299456
- [Background] Tan R, Cano L, Lago-Rodriguez A, Dominguez R. The Effects of Dietary Nitrate Supplementation on Explosive Exercise Performance: A Systematic Review. Int J Environ Res Public Health. 2022 Jan 11;19(2):762. doi: 10.3390/ijerph19020762. PMID 35055584
- [Background] Senefeld JW, Wiggins CC, Regimbal RJ, Dominelli PB, Baker SE, Joyner MJ. Ergogenic Effect of Nitrate Supplementation: A Systematic Review and Meta-analysis. Med Sci Sports Exerc. 2020 Oct;52(10):2250-2261. doi: 10.1249/MSS.0000000000002363. PMID 32936597
- [Background] Salem A, Ammar A, Kerkeni M, Boujelbane MA, Uyar AM, Kobel LM, Selvaraj S, Zare R, Heinrich KM, Jahrami H, Tounsi S, Zmijewski P, Schollhorn WI, Trabelsi K, Chtourou H. Short-Term Beetroot Juice Supplementation Enhances Strength, Reduces Fatigue, and Promotes Recovery in Physically Active Individuals: A Randomized, Double-Blind, Crossover Trial. Nutrients. 2025 May 19;17(10):1720. doi: 10.3390/nu17101720. PMID 40431460
- [Background] Murphy MJ, Rushing BR, Sumner SJ, Hackney AC. Dietary Supplements for Athletic Performance in Women: Beta-Alanine, Caffeine, and Nitrate. Int J Sport Nutr Exerc Metab. 2022 Feb 23;32(4):311-323. doi: 10.1123/ijsnem.2021-0176. Print 2022 Jul 1. PMID 35196646
- [Background] Miraftabi H, Avazpoor Z, Berjisian E, Sarshin A, Rezaei S, Dominguez R, Reale R, Franchini E, Samanipour MH, Koozehchian MS, Willems MET, Rafiei R, Naderi A. Effects of Beetroot Juice Supplementation on Cognitive Function, Aerobic and Anaerobic Performances of Trained Male Taekwondo Athletes: A Pilot Study. Int J Environ Res Public Health. 2021 Sep 28;18(19):10202. doi: 10.3390/ijerph181910202. PMID 34639501
- [Background] Lopez-Samanes A, Ramos-Alvarez JJ, Miguel-Tobal F, Gaos S, Jodra P, Arranz-Munoz R, Dominguez R, Montoya JJ. Influence of Beetroot Juice Ingestion on Neuromuscular Performance on Semi-Professional Female Rugby Players: A Randomized, Double-Blind, Placebo-Controlled Study. Foods. 2022 Nov 12;11(22):3614. doi: 10.3390/foods11223614. PMID 36429210
- [Background] Jones AM, Vanhatalo A, Seals DR, Rossman MJ, Piknova B, Jonvik KL. Dietary Nitrate and Nitric Oxide Metabolism: Mouth, Circulation, Skeletal Muscle, and Exercise Performance. Med Sci Sports Exerc. 2021 Feb 1;53(2):280-294. doi: 10.1249/MSS.0000000000002470. PMID 32735111
- [Background] Esen O, Karayigit R, Peart DJ. Acute beetroot juice supplementation did not enhance intermittent running performance in trained rugby players. Eur J Sport Sci. 2023 Dec;23(12):2321-2328. doi: 10.1080/17461391.2023.2230942. Epub 2023 Jul 13. PMID 37394944
- [Background] d'Unienville NMA, Blake HT, Coates AM, Hill AM, Nelson MJ, Buckley JD. Effect of food sources of nitrate, polyphenols, L-arginine and L-citrulline on endurance exercise performance: a systematic review and meta-analysis of randomised controlled trials. J Int Soc Sports Nutr. 2021 Dec 29;18(1):76. doi: 10.1186/s12970-021-00472-y. PMID 34965876
- [Background] Dominguez R, Mate-Munoz JL, Cuenca E, Garcia-Fernandez P, Mata-Ordonez F, Lozano-Estevan MC, Veiga-Herreros P, da Silva SF, Garnacho-Castano MV. Effects of beetroot juice supplementation on intermittent high-intensity exercise efforts. J Int Soc Sports Nutr. 2018 Jan 5;15:2. doi: 10.1186/s12970-017-0204-9. eCollection 2018. PMID 29311764
- [Background] Delleli S, Ouergui I, Messaoudi H, Trabelsi K, Glenn JM, Ammar A, Chtourou H. Does Beetroot Supplementation Improve Performance in Combat Sports Athletes? A Systematic Review of Randomized Controlled Trials. Nutrients. 2023 Jan 12;15(2):398. doi: 10.3390/nu15020398. PMID 36678270

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Following approval by the ethics committee, two rugby groups located in Bogotá, Colombia, were contacted. The project was explained, questions answered, and an invitation to participate was extended. Two weeks before the physical tests, an initial screening was conducted with those interested to verify compliance with inclusion and exclusion criteria. Informed consent was obtained. Instructions were also given, such as not using mouthwash and a list of nitrate-rich foods to avoid.
Pre-assignment Details: Before the assignment, a nutritional assessment was performed, verifying inclusion and exclusion criteria, as well as educating about the nitrate washout period and the use of mouthwash that may affect the research. Thus, it was recommended not to consume foods rich in nitrates from 3 days before the study until its completion. A list of these foods was provided and the requirement to not use mouthwash during the same period.
Period: Overall Study
Arm/Group | Placebo-Beetroot | Beetroot-Placebo
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The groups are distributed randomly, ensuring that there are both men and women.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo-Beetroot | Beetroot-Placebo | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 22.4 [20 to 24] | 25.6 [19 to 33] | 24 [20 to 25]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 2 | 3 | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Time training rugby [Mean (Standard Deviation); unit: years] | 2.8 (1.9) | 7.6 (4.8) | 5.2 (4.3)

OUTCOME MEASURES:

1. Primary Outcome: Results Obtained in the Physical Tests to Evaluate Impact on Acceleration
Description: Physical tests are performed over two different weeks. Initially, the 40-meter sprint test is performed with two attempts, with the attempt with the shortest execution time being considered. Distances from 0 to 10 meters are used to evaluate acceleration in meters per second squared (m/s^2)
Time Frame: First and second physical tests weeks
Measure: Mean (Inter-Quartile Range); unit: m/s^2
Groups:
- Placebo-Beetroot: The group receives the placebo the first week and the beetroot the second week.
  Placebo and Beetroot in the form of waffles to ensure the study is blinded.
  40 meters sprint: The participant performs a race at maximum speed with two attempts, times are taken at 10, 30 and 40 meters, to evaluate acceleration and speed, the attempt with the shortest times is the one taken for the research.
- Beetroot-Placebo: The group receives the beetroot the first week and the placebo the second week.
  Participants receive the beetroot and placebo in the form of waffles to ensure the study is blinded.
  40 meters sprint: The participant performs a race at maximum speed with two attempts, times are taken at 10, 30 and 40 meters, to evaluate acceleration and speed, the attempt with the shortest times is the one taken for the research.
Arm/Group | Placebo-Beetroot | Beetroot-Placebo
Number analyzed (Participants) | 5 | 5
m/s^2
  Placebo | 1.76 [1.64 to 2.01] | 2.44 [2.20 to 2.55]
  Beetroot | 2.08 [2.03 to 2.18] | 2.19 [1.59 to 2.31]
Statistical Analysis 1: Comparison: Placebo-Beetroot vs Beetroot-Placebo; Test type: Superiority; p = 0.8705, t-test, 2 sided; Mean Difference (Net) = 0.04 — Beetroot effect

2. Primary Outcome: Speed Results Over Distance From 0 to 30 Meters in 40 Meters Sprint Test
Description: In the 40-meter speed test, the time taken to travel from the start to the 30 meters is measured in meters per second (m/s)
Time Frame: First and second physical tests weeks
Measure: Mean (Inter-Quartile Range); unit: m/s
Arm/Group | Placebo-Beetroot | Beetroot-Placebo
Number analyzed (Participants) | 5 | 5
m/s
  Placebo | 5.61 [5.16 to 6.04] | 6.46 [5.87 to 6.73]
  Beetroot | 5.85 [5.44 to 6.38] | 6.25 [5.67 to 6.80]
Statistical Analysis 1: Comparison: Placebo-Beetroot vs Beetroot-Placebo; Test type: Superiority; p = 0.9161, t-test, 2 sided; Mean Difference (Net) = 0.01 — Beetroot effect

3. Primary Outcome: Maximum Speed Results With the Distance of 30 to 40 Meters in the 40-meter Sprint Test
Description: In the 40-meter sprint test, the time to cover from a distance of 30 meters to 40 meters is measured in meters per second (m/s)
Time Frame: First and second physical tests weeks
Measure: Mean (Inter-Quartile Range); unit: m/s
Arm/Group | Placebo-Beetroot | Beetroot-Placebo
Number analyzed (Participants) | 5 | 5
m/s
  Placebo | 7.74 [7.41 to 8.47] | 8.06 [7.75 to 8.55]
  Beetroot | 7.47 [6.33 to 7.81] | 8.02 [7.58 to 8.62]
Statistical Analysis 1: Comparison: Placebo-Beetroot vs Beetroot-Placebo; Test type: Superiority; p = 0.4166, t-test, 2 sided; Mean Difference (Net) = -0.15 — Beetroot effect

4. Primary Outcome: Speed Given by Distance From 0 to 40 Meters Sprint
Description: Time to cover the distance from 0 to 40 meters sprint at maximum speed in meters per second (m/s)
Time Frame: First and second physical tests weeks
Measure: Mean (Inter-Quartile Range); unit: m/s
Arm/Group | Placebo-Beetroot | Beetroot-Placebo
Number analyzed (Participants) | 5 | 5
m/s
  Placebo | 6.00 [5.47 to 6.50] | 6.78 [6.37 to 7.25]
  Beetroot | 6.17 [5.59 to 6.77] | 6.61 [6.14 to 7.25]
Statistical Analysis 1: Comparison: Placebo-Beetroot vs Beetroot-Placebo; Test type: Superiority; p = 0.9995, t-test, 2 sided; Mean Difference (Net) = 0 — Beetroot effect

5. Primary Outcome: Fitness Results From the Bronco Test
Description: Fitness is assessed by the time it takes to cover the 1.2 km Bronco test segmented into distances of 20, 40, and 60 meters, which are covered 5 times.
Time Frame: First and second physical tests weeks
Measure: Mean (Inter-Quartile Range); unit: Minutes
Groups:
- Placebo-Beetroot: The group receives the placebo the first week and the following week they receive the beetroot
  Participants receive the placebo and beetroot in the form of waffles to ensure the study is blinded, as the 6 mmol of nitrates used require a high concentration of beetroot, which is masked by the waffle ingredients and food coloring.
  Fitness test by bronco test: The participant runs a distance of 20, 40, and 60 meters, back and forth, 5 times at maximum speed. The variable to be measured is the total time taken to complete the test.
- Beetroot-Placebo: The group receives the beetroot the first week and the following week receives the placebo.
  Participants receive the placebo and beetroot in the form of waffles to ensure the study is blinded, as the 6 mmol of nitrates used require a high concentration of beetroot, which is masked by the waffle ingredients and food coloring.
  Fitness test by bronco test: The participant runs a distance of 20, 40, and 60 meters, back and forth, 5 times at maximum speed. The variable to be measured is the total time taken to complete the test.
Arm/Group | Placebo-Beetroot | Beetroot-Placebo
Number analyzed (Participants) | 5 | 5
Minutes
  Placebo | 6.08 [5.88 to 6.13] | 5.60 [5.38 to 5.78]
  Beetroot | 5.95 [5.72 to 6.07] | 5.54 [5.27 to 5.82]
Statistical Analysis 1: Comparison: Placebo-Beetroot vs Beetroot-Placebo; Test type: Superiority; p = 0.0422, t-test, 2 sided; Mean Difference (Net) = -0.09 — Beetroot effect

6. Primary Outcome: Maximum Strength in the Lower-body Given by Squat
Description: Squats are performed technically until reaching 1 repetition maximum (1RM) meeting technical requirements.
Time Frame: First and second physical tests weeks
Measure: Mean (Inter-Quartile Range); unit: kilograms (kg)
Groups:
- Placebo-Beetroot: The group receives the placebo the first week and the following week they receive the beetroot
  Participants receive the beetroot and placebo in the form of waffles to ensure the study is blinded, as the 6 mmol of nitrates used require a high concentration of beetroot, which is masked by the waffle ingredients and food coloring.
  Maximal strength: Each participant performs squats and bench press to evaluate lower-body and upper-body maximal strength, thus identifying their maximum strength taken per kilogram lifted.
- Beetroot-Placebo: The group receives the beetroot the first week and the following week receives the placebo.
  Participants receive the beetroot and placebo in the form of waffles to ensure the study is blinded, as the 6 mmol of nitrates used require a high concentration of beetroot, which is masked by the waffle ingredients and food coloring.
  Maximal strength: Each participant performs squats and bench press to evaluate lower-body and upper-body maximal strength, thus identifying their maximum strength taken per kilogram lifted.
Arm/Group | Placebo-Beetroot | Beetroot-Placebo
Number analyzed (Participants) | 4 | 5
kilograms (kg)
  Placebo | 101.25 [67.5 to 118.75] | 116.0 [85.0 to 130.0]
  Beetroot | 108.75 [73.75 to 127.50] | 120.0 [85.0 to 140.0]
Statistical Analysis 1: Comparison: Placebo-Beetroot vs Beetroot-Placebo; Test type: Superiority; p = 0.0027, t-test, 2 sided; Mean Difference (Net) = 5.56 — Beetroot effect

7. Primary Outcome: Maximum Upper-body Strength Given by Bench Press Test
Description: Maximum weight lifted in 1 maximum repetition in a technically correct manner in the bench press exercise
Time Frame: First and second physical tests weeks
Measure: Mean (Inter-Quartile Range); unit: kilograms (kg)
Arm/Group | Placebo-Beetroot | Beetroot-Placebo
Number analyzed (Participants) | 5 | 5
kilograms (kg)
  Placebo | 49.4 [30.0 to 55.0] | 72.2 [47.0 to 85.0]
  Beetroot | 52.8 [33.0 to 58.0] | 71.2 [45.0 to 82.0]
Statistical Analysis 1: Comparison: Placebo-Beetroot vs Beetroot-Placebo; Test type: Superiority; p = 0.2598, t-test, 2 sided; Mean Difference (Net) = 1.2 — Beetroot effect

8. Primary Outcome: Perception of Fatigue Given by the Borg Scale
Description: According to a score of 1 to 10, with 1 being the lowest and 10 being the highest level of fatigue, participants evaluated their perception at the end of the physical tests.
Time Frame: First and second weeks at the end of the physical tests
Measure: Mean (Inter-Quartile Range); unit: units on a scale from 1 to 10
Groups:
- Placebo-Beetroot: The group receives the placebo the first week and the following week they receive the beetroot
  Participants receive the beetroot and placebo in the form of waffles to ensure the study is blinded, as the 6 mmol of nitrates used require a high concentration of beetroot, which is masked by the waffle ingredients and food coloring.
  Borg scale: At the end of the tests, each participant is asked to evaluate their perception of fatigue by giving a number between 1 and 10, with 1 being the lowest level of fatigue and 10 being the highest.
- Beetroot-Placebo: The group receives the beetroot the first week and the following week receives the placebo.
  Participants receive the beetroot and placebo in the form of waffles to ensure the study is blinded, as the 6 mmol of nitrates used require a high concentration of beetroot, which is masked by the waffle ingredients and food coloring.
  Borg scale: At the end of the tests, each participant is asked to evaluate their perception of fatigue by giving a number between 1 and 10, with 1 being the lowest level of fatigue and 10 being the highest.
Arm/Group | Placebo-Beetroot | Beetroot-Placebo
Number analyzed (Participants) | 5 | 5
units on a scale from 1 to 10
  Placebo | 4.6 [4.0 to 5.0] | 5.0 [4.0 to 6.0]
  Beetroot | 4.8 [4.0 to 6.0] | 3.6 [2.0 to 4.0]
Statistical Analysis 1: Comparison: Placebo-Beetroot vs Beetroot-Placebo; Test type: Superiority; p = 0.1725, Wilcoxon (Mann-Whitney); Mean Difference (Net) = -0.6 — Beetroot effect

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: Participants have no risk of death because they were not provided with any risk doses of food. All-Cause Mortality and Serious Adverse Events were not monitored/assessed.
  Other adverse events monitored: During and at the end of the research, questions were asked about gastrointestinal effects with the consumption of placebo and/or beetroot, and no adverse effects were observed.
Arm/Group | Placebo-Beetroot | Beetroot-Placebo
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

LIMITATIONS AND CAVEATS:
Recruiting a sample size was difficult; there aren't many rugby players in Colombia, and personal schedules didn't fit the study. Furthermore, it's a sport prone to recurrent injuries due to its high impact, so several participants withdrew due to injuries unrelated to the study, limiting the sample size.

The speed tests were measured subjectively, although they were performed with trained individuals; it would have been better to use technology to achieve greater accuracy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-01-15): https://cdn.clinicaltrials.gov/large-docs/89/NCT07106489/Prot_SAP_000.pdf
  • Informed Consent Form (2025-01-15): https://cdn.clinicaltrials.gov/large-docs/89/NCT07106489/ICF_001.pdf